CLINICAL TRIAL: NCT04624204
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study of Pembrolizumab (MK-3475) in Combination With Concurrent Chemoradiation Therapy Followed by Pembrolizumab With or Without Olaparib (MK-7339), Compared to Concurrent Chemoradiation Therapy Alone in Participants With Newly Diagnosed Treatment-Naïve Limited-Stage Small Cell Lung Cancer (LS-SCLC)
Brief Title: Placebo-controlled, Study of Concurrent Chemoradiation Therapy With Pembrolizumab Followed by Pembrolizumab and Olaparib in Newly Diagnosed Treatment-Naïve Limited-Stage Small Cell Lung Cancer (LS-SCLC) (MK 7339-013/KEYLYNK-013)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7339-013; MK-7339-013 (Other: MSD Protocol Number); jRCT2031200296 (Registry Identifier: jRCT); 2023-504959-27-00 (Registry Identifier: EU CT); U1111-1290-4870 (Registry Identifier: UTN); 2019-003616-31 (EudraCT Number)
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Small Cell Lung Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Pembrolizumab; Olaparib
MeSH Terms: conditions — Small Cell Lung Carcinoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Sodium Chloride; olaparib; BID protein, human; Etoposide; Platinum

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A - Pembrolizumab 200 mg (Experimental): Participants will receive 4 cycles of standard-of-care chemotherapy (etoposide/platinum) plus pembrolizumab 200 mg every 3 weeks (Q3W) concurrently with standard thoracic radiotherapy, followed by 9 cycles of pembrolizumab 400 mg every 6 weeks (Q6W) plus olaparib matching placebo twice daily (BID) for 12 months or until specific discontinuation criteria are met.
  Interventions: Biological: Pembrolizumab 200 mg; Biological: Pembrolizumab 400 mg; Drug: Olaparib matching placebo; Drug: Etoposide 100 mg/m^2; Drug: Platinum, investigator's choice; Radiation: Standard Thoracic Radiotherapy; Radiation: Prophylactic Cranial Irradiation (PCI)
- Group B - Pembrolizumab 200 mg plus Olaparib 300 mg BID (Experimental): Participants will receive 4 cycles of standard-of-care chemotherapy (etoposide/platinum) plus pembrolizumab 200 mg Q3W concurrently with standard thoracic radiotherapy, followed by 9 cycles of pembrolizumab 400 mg Q6W plus olaparib 300 mg BID for 12 months or until specific discontinuation criteria are met.
  Interventions: Biological: Pembrolizumab 200 mg; Biological: Pembrolizumab 400 mg; Drug: Olaparib 300 mg BID; Drug: Etoposide 100 mg/m^2; Drug: Platinum, investigator's choice; Radiation: Standard Thoracic Radiotherapy; Radiation: Prophylactic Cranial Irradiation (PCI)
- Group C (Pembrolizumab and Olaparib Matching Placebos) (Placebo Comparator): Participants will receive 4 cycles of standard-of-care chemotherapy (etoposide/platinum) plus pembrolizumab placebo (saline) Q3W concurrently with standard thoracic radiotherapy, followed by 9 cycles of pembrolizumab placebo (saline) Q6W plus olaparib matching placebo for 12 months or until specific discontinuation criteria are met.
  Interventions: Drug: Pembrolizumab placebo (saline); Drug: Olaparib matching placebo; Drug: Etoposide 100 mg/m^2; Drug: Platinum, investigator's choice; Radiation: Standard Thoracic Radiotherapy; Radiation: Prophylactic Cranial Irradiation (PCI)

INTERVENTIONS:
Biological: Pembrolizumab 200 mg — Pembrolizumab 200 mg Q3W
  Other Names: MK-3475; KEYTRUDA®
  Arms: Group A - Pembrolizumab 200 mg; Group B - Pembrolizumab 200 mg plus Olaparib 300 mg BID
Biological: Pembrolizumab 400 mg — Pembrolizumab 400 mg Q6W
  Other Names: MK-3475; KEYTRUDA®
  Arms: Group A - Pembrolizumab 200 mg; Group B - Pembrolizumab 200 mg plus Olaparib 300 mg BID
Drug: Pembrolizumab placebo (saline) — Pembrolizumab placebo (saline) Q3W
  Arms: Group C (Pembrolizumab and Olaparib Matching Placebos)
Drug: Pembrolizumab placebo (saline) — Pembrolizumab placebo (saline) Q6W
  Arms: Group C (Pembrolizumab and Olaparib Matching Placebos)
Drug: Olaparib 300 mg BID — Olaparib 300 mg twice daily (BID)
  Other Names: MK-7339; LYNPARZA®
  Arms: Group B - Pembrolizumab 200 mg plus Olaparib 300 mg BID
Drug: Olaparib matching placebo — Olaparib matching placebo BID
  Arms: Group A - Pembrolizumab 200 mg; Group C (Pembrolizumab and Olaparib Matching Placebos)
Drug: Etoposide 100 mg/m^2 — Etoposide 100 mg/m^2 intravenous (IV) Q3W, Day 1-3
Drug: Platinum, investigator's choice — Carboplatin titrated to an area under the plasma drug concentration time curve (AUC) of 5 mg/mL/min IV Q3W OR Cisplatin 75 mg/m^2 IV Q3W on Day 1 of each cycle
Radiation: Standard Thoracic Radiotherapy — Standard Thoracic Radiotherapy
Radiation: Prophylactic Cranial Irradiation (PCI) — PCI will be strongly recommended for participants who achieve CR or PR after completion of chemoradiation treatment.

SUMMARY:
Researchers are looking for new ways to treat Limited-Stage Small Cell Lung Cancer (LS-SCLC), a type of lung cancer that has not spread from the lung to other parts of the body. The purpose of this study is to learn if pembrolizumab and olaparib, when given with chemotherapy and radiation treatment (CRT), can be effective in treating LS-SCLC. The researchers want to know if participants who receive CRT and pembrolizumab, with or without olaparib, have a longer overall survival compared to participants who only receive CRT.

ELIGIBILITY:
Inclusion Criteria:

1. Has pathologically (histologically or cytologically) confirmed Small Cell Lung Cancer (SCLC).

   Note: Note: Participants with histology showing a mixed tumor with small cell and non-small cell elements are not eligible.
2. Has Limited-Stage SCLC (Stage I-III, by AJCC 8th Edition Cancer Staging), and can be safely treated with definitive radiation doses.
3. Has no evidence of metastatic disease by whole body positron emission tomography /computed tomography (PET/CT scan), CT or magnetic resonance imaging (MRI) scans
4. Has at least 1 lesion that meets the criteria for being measurable, as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
5. Has not received prior treatment (chemotherapy or radiotherapy or surgery resection) of LS-SCLC.
6. Is not expected to require tumor resection during the course of the study.
7. Must submit a pre-treatment tumor tissue sample (formalin-fixed, paraffin embedded blocks are preferred to slides) including cytologic sample, if tissue sample unavailable.
8. Has Eastern Cooperative Oncology Group (ECOG) Performance score 0 or 1 assessed within 7 days prior to the first administration of study intervention.
9. Has a life expectancy of at least 6 months.
10. Has adequate organ function.
11. Male and female participants who are not pregnant and of childbearing potential must follow contraceptive guidance during the treatment period and for the time needed to eliminate each study intervention.
12. Male and female participants who are at least 18 years of age at the time of signing the information consent.
13. Male participants must refrain from donating sperm during the treatment period and for the time needed to eliminate each study intervention.
14. Abstains from breastfeeding during the study intervention period and for at least the following period after the last study intervention:

    * Pembrolizumab: 120 days
    * Olaparib: 7 days

Exclusion Criteria:

1. Has history, current diagnosis, or features suggestive of myelodysplastic syndrome/ acute myeloid leukemia (MDS/AML).
2. Has received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti-programmed cell death ligand 1 (anti-PDL1), or anti- programmed cell death ligand 2 (anti-PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor
3. Has received prior therapy with olaparib or with any other polyadenosine 5'diphosphoribose (polyADP ribose) polymerization (PARP) inhibitor.
4. Had major surgery <4 weeks prior to the first dose of study intervention (except for placement of vascular access).
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
8. Has severe hypersensitivity (≥ Grade 3) to study intervention and/or any of its excipients.
9. Has an active autoimmune disease that has required systemic treatment in past 2 years
10. Has a history of (non-infectious) pneumonitis/interstitial lung disease that requires steroids
11. Has an active infection requiring systemic therapy.
12. Has a known history of human immunodeficiency virus (HIV) infection or Hepatitis B or known active Hepatitis C virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1); the time from randomization to progression or death due to any cause, whichever occurs first | Up to approximately 59 months
  Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) is the time from randomization to progression or death due to any cause, whichever occurs first.
Overall Survival: the time from randomization to death due to any cause | Up to approximately 82 months
  Overall Survival (OS) is the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Number of Participants Experiencing an Adverse Events (AEs) | Up to approximately 82 months
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Number of Participants Discontinuing Study Treatment Due to Adverse Events (AEs) | Up to approximately 82 months
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Objective Response (OR): Complete Response (CR) or Partial Response (PR) | Up to approximately 82 months
  Percentage of participants in the analysis population who have a best overall response of either confirmed CR or a PR per RECIST 1.1.
Duration of Response (DOR): the time from the earliest date of first documented evidence of confirmed CR or PR until the earliest date of disease progression or death from any cause, whichever comes first | Up to approximately 82 months
  DOR is the time from the earliest date of first documented evidence of confirmed CR or PR until the earliest date of disease progression or death from any cause, whichever comes first.
Change from Baseline at Cycle 1 in European Organization for Research and Treatment (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status / Quality of Life (Items 29 & 30) Scale Score | Baseline and 82 months post randomization
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "How would you rate your overall health during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 scores will be presented.
Change from Baseline at Cycle 1 in EORTC Quality of Life Questionnaire Lung Cancer Module 13 (QLQ-LC13) Cough (Item 1) Scale Score | Baseline and 82 months post randomization
  The EORTC QLQ-LC13 is a lung cancer specific supplemental questionnaire used in combination with the EORTC QLQC30 questionnaire. Participant responses to the question "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. The change from baseline in EORTC QLQ-LC13 cough (Item 1) score will be presented.
Change from Baseline at Cycle 1 in EORTC QLQ-LC13 Chest Pain (Item 10) Scale Score | Baseline and 82 months post randomization
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQC30 questionnaire. Participant responses to the question "How was your chest pain?" are scored on a 4 point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. The change from baseline in EORTC QLQ-LC13 chest pain (Item 10) score will be presented.
Change from Baseline at Cycle 1 in EORTC QLQ-C30 Dyspnea (Item 8) Scale Score | Baseline and 82 months post randomization
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. The change from baseline in EORTC QLQ-LC13 dyspnea (Item 8) score will be presented.
Change from Baseline at Cycle 1 in EORTC QLQ-C30 Physical Functioning (Items 1 to 5) Scale Score | Baseline and 82 months post randomization
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better quality of life. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) score will be presented.
Time to True Deterioration (TTD) in EORTC QLQ-C30 Global Health Status / Quality of Life (Items 29 & 30) Scale Score | Up to approximately 82 months post randomization
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "How would you rate your overall health during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. TTD was defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in EORTC QLQ-C30 Items 29 and 30 scale scores.
Time to True Deterioration (TTD) in Cough (LC13/Item 1) Scale Score | Up to approximately 82 months post randomization
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQC30 questionnaire. Participant responses to the question "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. TTD was defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in cough EORTC QLQLC13 cough (Item 1) scale score.
Time to True Deterioration (TTD) in Chest Pain (LC13/Item 10) Scale Score | Up to approximately 82 months post randomization
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQC30 questionnaire. Participant responses to the question "How was your chest pain?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. TTD was defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in EORTC QLQ-LC13 chest pain (Item 10) scale score.
Time to True Deterioration (TTD) in EORTC QLQ-C30 Dyspnea (Item 8) Scale Score | Up to approximately 82 months post randomization
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. TTD was defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in EORTC QLQ-C30 dyspnea (Item 8) scale score.
Time to True Deterioration (TTD) in EORTC QLQ-C30 Physical Functioning (Items 1 to 5) Scale Score | Up to approximately 82 months post randomization
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better quality of life. TTD was defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in EORTC QLQ-C30 physical functioning (Items 1 to 5) scale scores.
Objective Response (OR, according to RECIST 1.1 by BICR) assessed by programmed cell death ligand 1 (PD-L1) expression levels | Up to approximately 82 months
  Percentage of participants in the analysis population who have a best overall response of either confirmed CR or a PR per RECIST 1.1, analyzed by programmed cell death ligand 1 (PD-L1) expression levels.
Duration of Response (DOR, according to RECIST 1.1 by BICR) assessed by programmed cell death ligand 1 (PD-L1) expression levels | Up to approximately 82 months
  DOR is the time from the earliest date of first documented evidence of confirmed CR or PR until the earliest date of disease progression or death from any cause, whichever comes first, analyzed by programmed cell death ligand 1 (PD-L1) expression levels.
Progression-free Survival (PFS, according to RECIST 1.1 by BICR) assessed by programmed cell death ligand 1 (PD-L1) expression levels | Up to approximately 59 months
  Progression-free Survival Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1); the time from randomization to progression or death due to any cause, whichever occurs first, analyzed by programmed cell death ligand 1 (PD-L1) expression levels.
Overall Survival (OS) assessed by programmed cell death ligand 1 (PD-L1) expression levels | Up to approximately 82 months
  Overall Survival: the time from randomization to death due to any cause, analyzed by programmed cell death ligand 1 (PD-L1) expression levels.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Merck Sharp & Dohme LLC
Locations (187):
- United States (35):
  - Ironwood Cancer & Research Centers ( Site 0007), Chandler, Arizona
  - Loma Linda University Cancer Center ( Site 0011), Loma Linda, California
  - Georgetown University ( Site 0017), Washington D.C., District of Columbia
  - Moffitt Cancer Center ( Site 0137), Tampa, Florida
  - University of Chicago Medical Center ( Site 0136), Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology ( Site 0034), Fort Wayne, Indiana
  - University of Kentucky Chandler Medical Center ( Site 0138), Lexington, Kentucky
  - Overton Brooks VAMC ( Site 0041), Shreveport, Louisiana
  - Harry & Jeanette Weinberg Cancer Institute ( Site 0045), Baltimore, Maryland
  - VA Ann Arbor Healthcare System ( Site 0050), Ann Arbor, Michigan
  - St. Vincent Healthcare Frontier Cancer Center ( Site 0056), Billings, Montana
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 0061), Omaha, Nebraska
  - Memorial Sloan Kettering - Basking Ridge ( Site 0133), Basking Ridge, New Jersey
  - John Theurer Cancer Center ( Site 0064), Hackensack, New Jersey
  - Memorial Sloan Kettering - Monmouth ( Site 0135), Middletown, New Jersey
  - Memorial Sloan Kettering - Bergen ( Site 0130), Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey ( Site 0123), New Brunswick, New Jersey
  - Memorial Sloan Kettering- Commack ( Site 0132), Commack, New York
  - Memorial Sloan Kettering - Westchester-Thoracic Oncology ( Site 0134), Harrison, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0069), New York, New York
  - Memorial Sloan Kettering - Nassau ( Site 0131), Uniondale, New York
  - Fairview Hospital-Moll Cancer Center ( Site 0141), Cleveland, Ohio
  - Cleveland Clinic Main ( Site 0139), Cleveland, Ohio
  - Cleveland Clinic - Hillcrest Hospital-Hillcrest Hospital Cancer Center ( Site 0140), Mayfield Heights, Ohio
  - Penn State Hershey Cancer Institute ( Site 0081), Hershey, Pennsylvania
  - Saint Francis Cancer Center ( Site 0087), Greenville, South Carolina
  - The University of Tennessee Medical Center ( Site 0116), Knoxville, Tennessee
  - Texas Oncology - Dallas (Presbyterian)_McIntyre ( Site 0098), Dallas, Texas
  - Texas Oncology - Dallas (Sammons) ( Site 0093), Dallas, Texas
  - MD Anderson Cancer Center ( Site 0100), Houston, Texas
  - Millennium Research & Clinical Development ( Site 0143), Houston, Texas
  - Providence Regional Cancer Partnership ( Site 0106), Everett, Washington
  - Medical Oncology Associates, PS ( Site 0142), Spokane, Washington
  - Multicare Institute For Research And Innovation ( Site 0108), Tacoma, Washington
  - Virginia Mason Memorial- North Star Lodge Cancer Center ( Site 0112), Yakima, Washington
- Australia (7):
  - Campbelltown Hospital ( Site 3002), Campbelltown, New South Wales
  - Nepean Hospital ( Site 3001), Kingswood, New South Wales
  - Calvary Mater Newcastle ( Site 3000), Waratah, New South Wales
  - Gold Coast University Hospital ( Site 3003), Southport, Queensland
  - Frankston Hospital-Oncology and Haematology ( Site 3007), Frankston, Victoria
  - Austin Health-Austin Hospital ( Site 3006), Heidelberg, Victoria
  - Western Health-Sunshine Hospital ( Site 3004), St Albans, Victoria
- Belgium (6):
  - Saint-Luc UCL ( Site 1005), Brussels, Bruxelles-Capitale, Region de
  - Grand Hopital de Charleroi ( Site 1003), Gilly, Hainaut
  - C.I.U. Hopital Ambroise Pare ( Site 1001), Mons, Hainaut
  - CHU UCL Namur Site de Godinne ( Site 1004), Yvoir, Namur
  - UZ Leuven ( Site 1002), Leuven, Vlaams-Brabant
  - AZ Delta ( Site 1000), Roeselare, West-Vlaanderen
- MHAT "Uni Hospital" OOD ( Site 2507), Panagyurishte, Pazardzhik, Bulgaria
- Canada (5):
  - Cross Cancer Institute ( Site 0206), Edmonton, Alberta
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0212), Hamilton, Ontario
  - CIUSSS Ouest de l Ile - St-Mary s Hospital ( Site 0202), Montreal, Quebec
  - McGill University Health Centre ( Site 0210), Montreal, Quebec
  - CIUSSS de la Mauricie et du Centre du Quebec ( Site 0200), Trois-Rivières, Quebec
- China (28):
  - Peking Union Medical College Hospital ( Site 3102), Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 3104), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Oncology Radiotherapy Department ( Site 3140), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 3127), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 3135), Chongqing, Chongqing Municipality
  - Daping Hospital,Third Military Medical University ( Site 3136), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 3126), Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 3121), Xiamen, Fujian
  - Peking University Shenzhen Hospital ( Site 3118), Shenzhen, Guangdong
  - Cancer Hospital Chinese Academy Of Medical Sciences. Shenzhen Center ( Site 3113), Shenzhen, Guangdong
  - Henan Cancer Hospital ( Site 3105), Zhengzhou, Henan
  - Tongji Medical College Huazhong University of Science and Technology ( Site 3138), Wuhan, Hubei
  - Union Hospital, Tongji Medical College of HUST ( Site 3123), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 3120), Wuhan, Hubei
  - Xiangya Hospital of Central South University ( Site 3137), Changsha, Hunan
  - Second Xiangya Hospital of Central-South University ( Site 3128), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 3133), Changsha, Hunan
  - Jiangsu Cancer Hospital ( Site 3139), Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University ( Site 3106), Nanchang, Jiangxi
  - The First Hospital of Jilin University ( Site 3132), Changchun, Jilin
  - Affiliated Cancer Hospital of Shandong First Medical University ( Site 3100), Jinan, Shandong
  - Shanghai Chest Hospital ( Site 3107), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital ( Site 3101), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University ( Site 3114), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital ( Site 3103), Tianjin, Tianjin Municipality
  - Hangzhou Cancer Hospital ( Site 3129), Hanghzou, Zhejiang
  - The 1st Affil Hosp of College of Medicine, Zhejiang Univ ( Site 3131), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 3108), Hangzhou, Zhejiang
- Estonia (2):
  - SA Pohja-Eesti Regionaalhaigla ( Site 2201), Tallinn, Harju
  - SA Tartu Ulikooli Kliinikum ( Site 2200), Tartu, Tartu
- France (9):
  - C.H. de Saint Quentin ( Site 1111), Saint-Quentin, Aisne
  - CHU de Bordeaux Hop St ANDRE ( Site 1115), Bordeaux, Aquitaine
  - Clinique Clairval ( Site 1108), Marseille, Bouches-du-Rhone
  - CHU Grenoble -Hop Michallon ( Site 1102), Grenoble, Isere
  - Institut De Cancerologie De L Ouest ( Site 1110), Saint-Herblain, Loire-Atlantique
  - Institut de Cancerologie de l Ouest Site Paul Papin ( Site 1103), Angers, Maine-et-Loire
  - Hopital Avicenne ( Site 1106), Bobigny, Seine-Saint-Denis
  - H.I.A. Sainte-Anne ( Site 1101), Toulon, Var
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 1105), Paris, Île-de-France Region
- Greece (5):
  - Henry Dunant Hospital ( Site 1205), Athens, Attica
  - Sotiria Regional Chest Diseases Hospital of Athens ( Site 1200), Athens, Attica
  - Anti-Cancer Hospital of Thessaloniki Theagenio ( Site 1204), Thessaloniki, Central Macedonia
  - University General Hospital of Herakleion ( Site 1202), Heraklion, Irakleio
  - University General Hospital of Larisa ( Site 1201), Larissa, Thessaly
- Hungary (6):
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 1306), Kecskemét, Bács-Kiskun county
  - Petz Aladar Megyei Oktato Korhaz ( Site 1312), Győr, Győr-Moson-Sopron
  - Reformatus Pulmonologiai Centrum ( Site 1304), Törökbálint, Pest County
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 1301), Budapest
  - Orszagos Onkologiai Intezet ( Site 1310), Budapest
  - Uzsoki Utcai Korhaz ( Site 1303), Budapest
- Israel (2):
  - Rambam Health Care Campus-Oncology Division ( Site 1401), Haifa
  - Chaim Sheba Medical Center ( Site 1400), Ramat Gan
- Italy (9):
  - A O U Policlinico di Modena ( Site 1503), Modena, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Careggi ( Site 1509), Florence, Firenze
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento-Oncology Unit ( Site 1513), Verona, Veneto
  - Azienda Ospedaliera Spedali Civili di Brescia ( Site 1512), Brescia
  - IRCCS Ospedale San Raffaele ( Site 1500), Milan
  - Istituto Nazionale dei Tumori ( Site 1504), Milan
  - Istituto Europeo di Oncologia ( Site 1501), Milan
  - IRCCS Istituto Oncologico Veneto ( Site 1506), Padua
  - Policlinico Universitario Agostino Gemelli ( Site 1505), Roma
- Japan (16):
  - Aichi Cancer Center ( Site 4010), Nagoya, Aichi-ken
  - Kobe Minimally Invasive Cancer Center ( Site 4003), Kobe, Hyōgo
  - Takarazuka City Hospital ( Site 4013), Takarazuka, Hyōgo
  - Kanagawa Cancer Center ( Site 4001), Yokohama, Kanagawa
  - Kansai Medical University Hospital ( Site 4009), Hirakata, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 4007), Takatsuki, Osaka
  - Shizuoka Cancer Center ( Site 4014), Nakatogari, Shizuoka
  - National Hospital Organization Kyushu Cancer Center ( Site 4000), Fukuoka
  - Niigata Cancer Center Hospital ( Site 4004), Niigata
  - Okayama University Hospital ( Site 4012), Okayama
  - Osaka International Cancer Institute ( Site 4005), Osaka
  - National Cancer Center Hospital ( Site 4015), Tokyo
  - Juntendo University Hospital ( Site 4008), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 4011), Tokyo
  - Cancer Institute Hospital of JFCR ( Site 4006), Tokyo
  - Showa Medical University Hospital ( Site 4002), Tokyo
- Lithuania (2):
  - Nacionalinis Vezio Institutas ( Site 2300), Vilnius, Vilniaus Miestas
  - LSMUL Kauno Klinikos ( Site 2301), Kaunas
- Mexico (2):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0401), Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" ( Site 0404), Monterrey, Nuevo León
- Portugal (3):
  - Unidade Local de Saude de Santa Maria - Hospital Pulido Valente ( Site 1704), Lisbon, Lisbon District
  - Inst. Portugues de Oncologia de Lisboa Francisco Gentil EPE ( Site 1705), Lisbon
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil E.P.E. ( Site 1701), Porto
- Romania (5):
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 2803), Cluj-Napoca, Cluj
  - Amethyst Radiotherapy Center-Oncologie Medicala ( Site 2805), Florești, Cluj
  - Spitalul Municipal Ploiesti ( Site 2801), Ploieşti, Prahova
  - Cabinet Medical Oncomed ( Site 2802), Timișoara, Timiș County
  - S.C.Focus Lab Plus S.R.L ( Site 2804), Bucharest
- Russia (7):
  - Main Military Clinical Hospital n.a. N.N.Burdenko ( Site 1812), Moscow, Moscow
  - MROI n.a. P.A. Herzen - branch of FSBI NMICR of MoH of Russia ( Site 1800), Moscow, Moscow
  - Moscow Regional Oncological Dispensary-Oncology (thoracic surgery) Department №1 ( Site 1815), Balashikha, Moscow Oblast
  - Nizhniy Novgorod Region Oncology Dispensary ( Site 1811), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Omsk Clinical Oncology Dispensary ( Site 1806), Omsk, Omsk Oblast
  - Sverdlovsk Regional Oncology Hospital ( Site 1807), Yekaterinburg, Sverdlovsk Oblast
  - Republican Clinical Oncology Dispensary-Chemotherapy #1 ( Site 1814), Kazan', Tatarstan, Respublika
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia ( Site 2995), Belgrade, Beograd
  - Institut za plucne bolesti Vojvodine Sremska Kamenica ( Site 2991), Kamenitz, Sremski Okrug
- South Africa (2):
  - Steve Biko Academic Hospital ( Site 5000), Pretoria, Gauteng
  - Groote Schuur Hospital ( Site 5002), Cape Town, Western Cape
- South Korea (8):
  - National Cancer Center ( Site 3306), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 3301), Seongnam-si, Kyonggi-do
  - The Catholic University of Korea St. Vincent s Hospital ( Site 3303), Suwon, Kyonggi-do
  - Inje University Haeundae Paik Hospital ( Site 3307), Busan, Pusan-Kwangyokshi
  - Asan Medical Center ( Site 3308), Songpagu, Seoul
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 3302), Daegu, Taegu-Kwangyokshi
  - Severance Hospital Yonsei University Health System ( Site 3304), Seoul
  - Samsung Medical Center ( Site 3300), Seoul
- Spain (6):
  - Hospital Duran i Reynals ( Site 1903), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Central de Asturias ( Site 1900), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d Hebron ( Site 1904), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 1902), Madrid
  - Hospital Regional Universitario de Malaga ( Site 1905), Málaga
  - Hospital Universitario Virgen Macarena-Unidad de Investigación Oncológica ( Site 1907), Seville
- Turkey (Türkiye) (5):
  - Ankara Bilkent Sehir Hastanesi ( Site 2007), Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 2009), Istanbul
  - Medipol Universite Hastanesi ( Site 2005), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 2003), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 2001), Izmir
- Ukraine (8):
  - Grigoriev Institute for medical Radiology NAMS of Ukraine ( Site 2110), Kharkiv, Kharkivs’ka Oblast’
  - Municipal non-profit Enterprise "Khmelnytskyi Regional Antitumor Center" ( Site 2115), Khmelnytskyi, Khmelnytskyi Oblast
  - LISOD. Hospital ( Site 2111), Pliuty, Kyiv Oblast
  - Medical Center of Yuriy Spizhenko LLC.-Clinical Trial ( Site 2104), Kapitanivka Village, Kyivska Oblast
  - Clinic of National Cancer Institute ( Site 2101), Kyiv, Kyivska Oblast
  - Medical Center Verum ( Site 2106), Kyiv, Kyivska Oblast
  - Communal Noncommercial Enterprise "Podillia Regional Oncolog-Chemotherapy Department ( Site 2114), Vinnytsia, Vinnytsia Oblast
  - Kyiv City Clinical Oncology Center ( Site 2100), Kyiv
- United Kingdom (6):
  - Royal Infirmary Aberdeen ( Site 2403), Aberdeen, Aberdeen City
  - Ninewells Hospital and Medical School ( Site 2401), Dundee, Dundee City
  - Taunton and Somerset Hospital ( Site 2404), Taunton, England
  - Barts Health NHS Trust ( Site 2409), London, London, City of
  - Guy s & St Thomas NHS Foundation Trust ( Site 2408), London, London, City of
  - The Christie NHS Foundation Trust ( Site 2405), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Rimner A, Lai WV, Califano R, Jabbour SK, Rudin CM, Faivre-Finn C, Cho BC, Kato T, Yu J, Chafin W, Yu L, Zhao B, Byers L. Rationale and Design of the Phase 3 KEYLYNK-013 Study of Pembrolizumab With Concurrent Chemoradiotherapy Followed by Pembrolizumab With or Without Olaparib for Limited-Stage Small-Cell Lung Cancer. Clin Lung Cancer. 2022 Jul;23(5):e325-e329. doi: 10.1016/j.cllc.2022.04.005. Epub 2022 Apr 29. PMID 35613997
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26265&tenant=MT_MSD_9011